CLINICAL TRIAL: NCT00738907
Title: Assessment of Beta Cell Mass by PET Scans With [11C] DTBZ in Longstanding Type 1 Diabetes
Brief Title: Assessment of Beta Cell Mass by PET Scans With [11C] Dihydrotetrabenazine (DTBZ) in Longstanding Type 1 Diabetes.
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paul Harris, Research Scientist, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Other Study IDs: DK77493 (completed)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2011-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We hypothesize that quantitative measurements of the beta cell mass within the endocrine pancreas can be obtained by PET via targeting of vesicular monoamine type 2 transporters with the radioligand [11C]DTBZ. and that there will be significant differences in [11C]DTBZ uptake in the anatomical space of the pancreas between normal individuals and those with BCM predicted to be greater or less than normal based on the measurement of insulin secretion.

DETAILED DESCRIPTION:
Diabetes results when the insulin secretory capacity of the beta cell population is lost or severely compromised. Plasma insulin levels have been used as a surrogate marker of beta cell mass (BCM) but insulin levels often do not correlate well with BCM and a "gold standard of measurement" to obtain this type of information would be of great value. The aim of the proposed study is to evaluate an islet imaging technique using PET scanning that will be able to be used for directly measuring BCM and thus provide valuable information for monitoring disease progress and response to therapy in people with diabetes and in people at high risk for diabetes. Type 1 diabetes (T1DM) occurs when the beta cells are selectively destroyed by a T cell mediated autoimmune process. People at high risk for developing T1DM, such as first degree relatives of patients with T1DM, can be sometimes be identified before the disease develops by measuring autoantibodies to beta cells, however this test is neither very sensitive or specific. In contrast, type 2 diabetes (T2DM) occurs in a setting of insulin resistance leading to hyperinsulinemia. In people at high risk for T2DM, beta cell mass increases to meet the demand for more insulin. The individual becomes diabetic when the BCM and insulin production can no longer compensate for the increased need for insulin, and blood glucose begins to rise. Loss of BCM may then occur as T2DM advances. People at high risk for T2DM include first degree relatives of patients with T2DM and those with obesity, insulin resistance and the metabolic syndrome. Little is known about the natural history of BCM, turnover and cell lifetime, or the course of inflammation in diabetes. This is principally because the pancreas is a highly heterogeneous organ that is difficult to biopsy without significant complications, and BCM is only 1-2% of the organ. Accurate assessment of BCM in human diabetes is limited to autopsy studies, which usually suffer from inadequate clinical information; thus, the development of noninvasive means of BCM measurement could be important, not only in intervention therapy of T1DM and T2DM, islet regeneration/stem cell therapy and islet transplantation.

Until recently, islet cell mass visualization has not been clinically feasible. We have previously identified a specific marker on pancreatic beta cells called vesicular monoamine transporter type 2 (VMAT2). In preclinical studies, we have shown that imaging beta cell mass with PET scanning using this radioligand is feasible in rats and in dosimetry studies conducted in baboons. This radioligand, [11C]DTBZ, has been used previously in human subjects in clinical trials evaluating P.E.T scanning of the brain in patients with bipolar illness and schizophrenia compared to healthy control subjects. In the current protocol, we propose to use a radioligand, [11C]DTBZ, that binds to VMAT2 in positron emission tomography (PET) scanning to assess whether PET can measure beta cell mass in human subjects.

ELIGIBILITY:
Inclusion Criteria: Potential participants must meet all of the following inclusion criteria:

1. Informed consent obtained from participants
2. Age 18 45 years
3. Healthy nondiabetic subjects will have normal fasting blood sugar (<100 mg/dl), BMI 18.5 24.9, no history of type 2 diabetes in first degree relative
4. Type 1 diabetes defined by: ADA criteria or judgment of physician; diabetes onset younger than age 18, duration >5 years, BMI 18.5 24.9. Insulin dose <0.8 units/kg/day. Fasting c-peptide < 0.1 ng/ml
5. Obese hyperinsulinemic subjects will have BMI > 30 and fasting insulin>20 and c-peptide> 4.6 ng/ml and normal fasting blood sugar <100 mg/dl.
6. Able to tolerate PET imaging: not claustrophobic, able to lie supine for 1.5 hours
7. Normal liver and renal function tests including normal spot urine microalbumin/creatinine; normal complete blood count (CBC) including hematocrit >31.8% in women, >36.7% in men, white blood cell count (WBC) >3.4 K/mm3 and platelet count >162 K/mm3
8. Adequate collateral circulation in the wrist as assessed by Allen Test.

Exclusion Criteria: Potential participants must not have any of the following exclusion criteria:

1. Previous or current treatment with drugs influencing beta cell function or insulin sensitivity (e.g. oral hypoglycemic agents, glucocorticoids); or with antipsychotic, antianxiety, or antidepressant medications (eg monoamine oxidase (MAO) inhibitors, 5HT inhibitors, tricyclic antidepressants); or treatment with reserpine; or treatment with beta2receptor agonists (eg, terbutaline); or treatment with anticoagulant medication.
2. History of movement disorder such as Parkinson's Disease or Huntington's Disease
3. History of or psychiatric illness such as depression, bipolar disease, anxiety or schizophrenia.
4. If a female of childbearing age, currently pregnant, breastfeeding or not using a form of birth control
5. Previous or current use of cocaine, methamphetamine, ecstasy ( 3,4 methylenedioxymethamphetamine (MDMA))
6. Current daily intake of caffeine >500 mg/day (>45 cups of coffee; >10 12oz cans of soda)
7. Current history of cigarette smoking
8. Consumption of more than 1 alcoholic drink per day
9. Evidence of chronic infection
10. History of malignancy
11. Any prior participation in other research protocols within the past year that involve radiation, with the exception of plain radiography studies (i.e., chest xrays).
12. Medical implant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pancreatic tracer binding as standardized uptake value (SUV) or binding potential (BPnd) | measured over 60-120 minutes
  Reflects tissue density of biomarker

CONTACTS AND LOCATIONS:
Overall Officials: PAUL HARRIS, PH.D, Principal Investigator — Columbia University

REFERENCES:
- See also: Results of study — http://www.ncbi.nlm.nih.gov/pubmed/19223416